CLINICAL TRIAL: NCT01877460
Title: The Effects of Isovolumetric Preloads of Sodium Alginate-enriched Chocolate Milk on Glycemia, Subjective Appetite and Food Intake in Healthy Young Men
Brief Title: Sodium Alginate in Chocolate Milk, Satiety and Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 26942
Record Dates: First submitted 2013-06-06; First posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Health; Appetite Regulation; Glucose Metabolism
Keywords: sodium alginate; chocolate milk; satiety; energy intake; glycemia; insulinemia
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sodium alginate-free chocolate milk (Experimental): Sodium alginate-free chocolate milk (1% fat) (Beatrice Ltd., Toronto, Ontario)
  Interventions: Other: Dietary intervention
- 1.25% sodium alginate chocolate milk (Experimental): Chocolate milk (Beatrice Ltd., Toronto, Ontario) with 1.25% sodium alginate
  Interventions: Other: Dietary intervention
- 2.5% sodium alginate chocolate milk (Experimental): Chocolate milk (Beatrice Ltd., Toronto, Ontario) with 2.5% sodium alginate
  Interventions: Other: Dietary intervention
- 2.5% sodium alginate milk-free water-based solution (Experimental): Water solution with 2.5% sodium alginate
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — All arms were given to all participants, in a randomized order, to be consumed within 10 min after 12-h overnight fasting.

SUMMARY:
This study compares the effects of isovolumetric (325 ml) preloads of chocolate milk supplemented with sodium alginates at incremental doses on inter-meal glucose levels, appetite scores and food intake in healthy adult men. The findings of this study will illustrate whether the addition of sodium alginate to chocolate milk will improve the glycemic properties of chocolate milk and will potentiate its satiating characteristics. This study will also elucidate whether sodium alginates, incorporated into chocolate milk, will influence glycemia, appetite sensations and food intake in a dose-dependent manner. It is hypothesized that there will be a synergy between milk and sodium alginate beyond either alone. When combined with milk components, sodium alginate is expected to improve glycemia and induce satiety more than does either milk alone or alginate alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* non-smoking male subjects,
* aged 20-30 years with a body mass index between 20 and 24.9 kg/m2, were recruited.

Exclusion Criteria:

* Breakfast skippers,
* smokers,
* dieters,
* individuals with lactose-intolerance or
* who are allergic to milk,
* individuals with gastrointestinal problems and
* individuals with diabetes or other metabolic diseases were excluded from the study.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Satiety Change | 0, 10, 20, 30, 45, 60, 75, 90 and 120 min (pre-meal) and 140, 170, 200, 230 and 260 min (post-meal) after consumption of the treatments
  Pre-meal changes from 0 min; Post-meal changes from 120 min
  Satiety scores (mm) were assessed using 100-mm "Motivation to Eat" visual analog scale questionnaires. A composite score of the four appetite questions, including Desire to Eat, Hunger, Fullness and Prospective Food Consumption, in the "Motivation to Eat" visual analog scale was calculated to obtain the average appetite score for statistical analysis.

SECONDARY OUTCOMES:
Food Intake | 120 min
  Food intake (kCal) was assessed 120 min after consumption of the treatments, using an ad libitum pizza lunch meal. Participants were asked to eat, during a 20-min period, until feeling comfortably full.

OTHER OUTCOMES:
Blood Glucose Change | 0, 10, 20, 30, 45, 60, 75, 90 and 120 min (pre-meal) and 140, 170, 200, 230 and 260 min (post-meal) after consumption of the treatments
  Pre-meal changes from 0 min; Post-meal changes from 120 min
  Blood glucose (mmol/L) was measured using finger prick capillary blood sample.
Serum Insulin Change | 0, 30, 60, 120 (pre-meal), and 140, 170 and 200 min (post-meal) after consumption of treatments
  Pre-meal changes from 0 min; Post-meal changes from 120 min
  Serum insulin (μU/mL) was measured using finger prick capillary blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, FitzGerald Building, Toronto, Ontario, Canada